CLINICAL TRIAL: NCT00341640
Title: Pharmacokinetics of Nicotine and Cotinine in Pregnant African-American Women and Implications for Pharmacological Interventions
Brief Title: Metabolism of Nicotine and Cotinine in Pregnant African-American Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999905074; 05-CH-N074
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-12-01

CONDITIONS: Pregnancy; Smokers
Keywords: Teen Pregnancy
MeSH Terms: interventions — Hematologic Tests

INTERVENTIONS:
Procedure: Blood testing

SUMMARY:
This study will provide information regarding the optimal dose and duration of nicotine replacement using the nicotine patch for a smoking cessation study of pregnant African-American women. Previous studies have shown that pregnancy, race and ethnicity can affect the way people metabolize nicotine. The information from this study may help scientists develop ways to help pregnant African-American women quit smoking and not start smoking again after delivery.

African-American women 18-30years of age who are in the second trimester of a healthy pregnancy, who are carrying only one baby and who smoke 10 or more cigarettes a day may be eligible for this study. Candidates are screened with a medical history, physical examination and urine test. They receive counseling to help them quit smoking. Those who cannot quit smoking within 7 to 10 days after receiving counseling may be invited to join the study.

Participants are admitted to a private room in the Pediatric Clinical Research Center at Children's National Medical Center in Washington, D.C., for 48 hours, during which time they are not permitted to smoke. After a "wash out" period, a nicotine patch will be applied according to these doses and schedules:

* 21 mg patch for 24 hours
* 21 mg patch for 16 hours
* 14 mg patch for 24 hours
* 14 mg patch for 16 hours

An intravenous (IV) line is placed in the subject's arm and 12 blood samples are drawn through the line at intervals during the 48 hours. Twleve urine and saliva samples are also collected. Blood, urine, and saliva samples are analyzed for nicotine and cotinine (a product of nicotine metabolism) levels, and DNA will be collected studied for genes that are associated with nicotine and cotinine metabolism. Participants are interviewed about their urges to smoke, quality of sleep, etc.

DETAILED DESCRIPTION:
This is a two-part protocol. This protocol is for Part A, the specific aims of which are to:

1. Determine the optimal dose (21 mg or 14 mg) and duration (24 hours or 16 hours) of nicotine replacement using the nicotine transdermal delivery device for African-American pregnant women who smoke, and
2. Determine the implications of the nicotine replacement studies for treatment with the nicotine replacement patch of African-American women who smoke during pregnancy.

Additional aims are to:

1. Collect DNA for exploratory analyses regarding genetic causes of differences in metabolism of nicotine and cotinine.

Latina/Hispanic women will not be included in this study because a) few smoke, and b) few are seen in the clinical sites from which participants will be recruited.

ELIGIBILITY:
* INCLUSION CRITERIA:

English-speaking, self-identified African-American women smokers, age 18 to 30 years, with singleton, uncomplicated pregnancies in the second trimester will be eligible.

Only women receiving routine prenatal care, begun by 16 weeks gestation, will be included.

Women will be asked to release records of their pregnancy to study staff for review prior to enrollment.

All participating women will receive clearance from their obstetrician before enrollment.

EXCLUSION CRITERIA:

Women who report use of any other substance of abuse besides nicotine will be ineligible.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Start 2005-01-06; Study Completion 2006-12-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Eskenazi B, Prehn AW, Christianson RE. Passive and active maternal smoking as measured by serum cotinine: the effect on birthweight. Am J Public Health. 1995 Mar;85(3):395-8. doi: 10.2105/ajph.85.3.395. PMID 7892926